CLINICAL TRIAL: NCT00970320
Title: Prevalence and Treatment of Anal Incontinence in Primiparous Women
Brief Title: Prevalence and Treatment of Anal Incontinence (AI) in Primiparous Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ostfold Hospital Trust (Other)
Collaborators: St. Olavs Hospital (Other); Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 3170
Record Dates: First submitted 2009-09-01; First posted 2009-09-02 (Estimated); Results first posted 2016-10-18 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-08

CONDITIONS: Fecal Incontinence
Keywords: Anal Incontinence; urinary incontinence; primiparas; prevalence; pelvic floor exercise treatment; Quality of Life (QoL)
MeSH Terms: conditions — Fecal Incontinence; Encopresis; Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Control group, RCT2 (No Intervention): Participants reporting anal incontinence 6 months postpartum receiving written information only for 6 months. After 6 months they are offered the same intervention as the intervention group, i.e. PFMT for 6 months.
- Intervention group, RCT 2 (Active Comparator): Participants reporting anal incontinence 6 months postpartum receiving pelvic floor muscle training (PFMT) for 6 months (+6 months).
  Interventions: Other: Pelvic floor muscle training
- Control group, RCT3 (No Intervention): Women with obsteric anal sphincter injury receiving written information only for 6 months. After 6 months they are offered the same intervention as the intervention group, i.e. PFMT for 6 months.
- Intervention group, RCT 3 (Active Comparator): Women with obsteric anal sphincter injury receiving pelvic floor muscle training (PFMT) for 6 months (+6 months).
  Interventions: Other: Pelvic floor muscle training
- Prevalence Study (No Intervention): 1571 primiparae delivering at Ostfold Hospital Trust or St. Olav's Hospital during the period May 2009 to December 2010.

INTERVENTIONS:
Other: Pelvic floor muscle training — 6 months of daily pelvic floor exercise treatment with regular follow up by specialist physiotherapist.
  Arms: Intervention group, RCT 2; Intervention group, RCT 3

SUMMARY:
Traumatic tears of the sphincter ani muscles after delivery may result in symptomatic urinary and anal incontinence, particularly in primiparas.

The efficacy of pelvic floor muscle exercise (PFME) in treating urinary incontinence (UI)is well documented, however, to date there is little evidence to support the efficacy of PFME in treating symptomatic anal incontinence.

This project consists of three separate studies. The prevalence survey/ study (1), investigates the prevalence of symptomatic anal incontinence among primiparas at Ostfold Hospital Trust Fredrikstad, Norway and St Olav's Hospital, Trondheim University Hospital, Norway, and the results in this study will form the basis of the two identical randomized controlled trials (RCT) investigating the treatment efficacy of PFME two groups of postpartum women. Women reporting symptomatic anal incontinence at six months postpartum (2) and women who have sustained a traumatic 3rd or 4th degree tear of the sphincter ani muscles during delivery (3), respectively, are randomized to an intervention group receiving PFME treatment for six months, or a control group. All RCT participants will undergo examination of PFM strength and activity, as well as anal ultrasound prior to randomization and after the intervention period.

DETAILED DESCRIPTION:
The recruitment in RCT ( 2) has been lower than expected (49/72). Due to financial reasons and problems with logistics and preparations for the main hospital (Ostfold Hospital Trust) moving into a new hospital, we were unable to extend the recruitment period in study 1. In RCT (3) AI was not an inclusion criterion. However, as both RCTs had the same outcome measure; anal incontinence, and a joint randomization process, stratified on hospital site and whether the participants had sustained an obsteric anal sphincter injury at delivery or not, the results from these studies will be reported together.

ELIGIBILITY:
Inclusion Criteria:

* primiparas aged 18 years or over with adequate knowledge of the Norwegian Language (prevalence study)
* Primiparas (Prevalence study and RCT 2)
* Women with obstetric anal sphincter injury with primary repair at delivery (RCT 3)

Exclusion Criteria all studies:

* Inadequate knowledge of the Norwegian language
* Diabetes mellitus
* Irritable bowel syndrome
* Neurological diseases such as Multiple Sclerosis
* Previous abdominal/colon surgery

In RCT studies:

Women who have already started pelvic floor muscle training postpartum due to severe anal incontinence or pelvic floor dysfunction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1718 (Actual)
Dates: Start 2009-05; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arvid Stordahl, MD PhD, Principal Investigator — Ostfold Hospital Trust
Locations (1):
- Ostfold Hospital Trust, Sarpsborg, Østfold fylke, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Johannessen HH, Wibe A, Stordahl A, Sandvik L, Backe B, Morkved S. Prevalence and predictors of anal incontinence during pregnancy and 1 year after delivery: a prospective cohort study. BJOG. 2014 Feb;121(3):269-79. doi: 10.1111/1471-0528.12438. Epub 2013 Sep 10. PMID 24021090
- [Result] Johannessen HH, Morkved S, Stordahl A, Sandvik L, Wibe A. Anal incontinence and Quality of Life in late pregnancy: a cross-sectional study. BJOG. 2014 Jul;121(8):978-87. doi: 10.1111/1471-0528.12643. Epub 2014 Mar 4. PMID 24589074
- [Result] Johannessen HH, Wibe A, Stordahl A, Sandvik L, Morkved S. Anal incontinence among first time mothers - what happens in pregnancy and the first year after delivery? Acta Obstet Gynecol Scand. 2015 Sep;94(9):1005-13. doi: 10.1111/aogs.12689. Epub 2015 Jun 23. PMID 26052628

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Primiparas during the period May 2009 and December 2010 and women sustaining obstetric anal sphincter injuries during the period 2009 to 2011 at Ostfold Hospital Trust and St. Olav's Hospital were invited to participate in the prevalence and intervention studies, respectively.
Groups:
- Prevalence Study: 1571 primiparas delivering at Ostfold Hospital Trust or St. Olav's Hospital during the period May 2009 to December 2010.
Period: Overall Study
Arm/Group | Control Group, RCT2 | Intervention Group, RCT 2 | Control Group, RCT3 | Intervention Group, RCT 3 | Prevalence Study
Started | 25 | 24 | 48 | 50 | 1571
Completed | 25 | 13 | 35 | 36 | 1031
Not Completed | 0 | 11 | 13 | 14 | 540

BASELINE CHARACTERISTICS:
Groups:
- Prevalence Study: 1571 primiparas delivering at Ostfold Hospital Trust or St. Olavs Hospital during the period May 2009 to December 2010.
- Total: Total of all reporting groups
Arm/Group | Control Group, RCT2 | Intervention Group, RCT 2 | Control Group, RCT3 | Intervention Group, RCT 3 | Prevalence Study | Total
Number analyzed (Participants) | 25 | 24 | 48 | 50 | 1571 | 1718
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 24 | 48 | 50 | 1571 | 1718
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.1 (3.9) | 27.8 (4.1) | 30.8 (4) | 30.5 (3.7) | 28.2 (4.7) | 29.3 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 24 | 48 | 50 | 1571 | 1718
  Male | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Norway | 25 | 24 | 48 | 50 | 1571 | 1718
Anal incontinence (AI) [Mean (Standard Deviation); unit: units on a scale] — The St Mark's score ranges from 0-24 points and measures the frequency of AI complaints. There is no standard grading of the scale. A change of +/- 5 points has been suggested as a minimal clinical important difference in severe AI patients, and +/- 2-3 points in less severely affected populations.
  units on a scale | 4.3 (4.0) | 4.5 (3.2) | 3.6 (3.3) | 4.1 (4.1) | 6.0 (5.0) | 4.5 (3.9)

OUTCOME MEASURES:

1. Primary Outcome: Change in Anal Incontinence as Measured on the St. Mark's Score
Description: Survey and interview using the questionnaire St. Mark's incontinence score ranging from 0 (no incontinence) -24 (complete incontinence) points for measuring anal incontinence (AI). The A total of 1069 women responded to the questionnaires at 6 months postpartum and 1031 at 12 months postpartum. Discrepancies in the number of included and analysed participants in the PFME trials are related to the number of women who did not attend the follow-up appointments as described in the published paper.
Time Frame: 0 to 24 months postpartum
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Prevalence Study: 1571 primiparae delivering at Ostfold Hospital Trust or St. Olavs Hospital during the period May 2009 to December 2010.
Arm/Group | Control Group, RCT2 | Intervention Group, RCT 2 | Control Group, RCT3 | Intervention Group, RCT 3 | Prevalence Study
Number analyzed (Participants) | 20 | 18 | 35 | 36 | 1571
units on a scale | 4.3 (4.0) | 4.5 (3.2) | 3.6 (3.3) | 4.1 (4.1) | 6.0 (5.0)

2. Secondary Outcome: Change in Urinary Incontinence as Measured on ICI-Q UI SF
Description: International Consultation of Incontinence Questionnaire, short form (ICI-Q SF) ranges from 0 (Complete continence) to 21 (Complete incontinence) and measures the frequency of UI, amount of leakage and impact on quality of life.
  Data have not been analysed.
Time Frame: 0 to 24 months postpartum
Reporting Status: Not Posted

3. Secondary Outcome: Fecal Incontinence of Life (FIQL) Scale
Description: Change in health-related quality of Life as measured on the fecal incontinence quality of life scale (FIQL). There is no total scale, only four sub scales ranging from 4 (complete continence, no impact on QoL) to 1 (complete incontinence, severe impact on QoL) Data from the postpartum period has not and will not be analysed due to low numbers.
Time Frame: 0 to 24 months postpartum
Reporting Status: Not Posted

4. Secondary Outcome: Change in Pelvic Floor Muscle Function Test as Measured on the ICS Scale
Description: Digital palpation and grading of voluntary pelvic floor muscle contraction (1=absent, 2=weak, 3=normal, 4=strong).
Time Frame: 12 to 24 months postpartum
Reporting Status: Not Posted

5. Secondary Outcome: Change in Manometry Measurements
Description: manometric measurements of pelvic floor muscle strength and anal sphincter length during voluntary pelvic floor muscle contraction
Time Frame: 12 to 24 months postpartum
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Throughout the studyperiod from 2009 to 2013
Description: no adverse events were registered during the study period
Arm/Group | Control Group, RCT2 | Intervention Group, RCT 2 | Control Group, RCT3 | Intervention Group, RCT 3 | Prevalence Study
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/24 | 0/48 | 0/50 | 0/1571
Other Adverse Events (participants affected / at risk) | 0/25 | 0/24 | 0/48 | 0/50 | 0/1571

LIMITATIONS AND CAVEATS:
Due to financial restrictions and Ostfold Hospital moving to a new hospital, the number of included participants were not as high as expected in RCT 2.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes